CLINICAL TRIAL: NCT03204929
Title: A Phase 1 Dose Escalation Study of Cu(II)ATSM Administered Orally to Patients With Early Idiopathic Parkinson's Disease
Brief Title: Dose Escalation Study of Cu(II)ATSM in Parkinson's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Collaborative Medicinal Development Pty Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMD-2016-002
Record Dates: First submitted 2017-06-28; First posted 2017-07-02 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — copper (II) diacetyl-di(N(4)-methylthiosemicarbazone); Copper

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Cu(II)ATSM (Experimental): Cu(II)ATSM dosed once daily
  Interventions: Drug: Cu(II)ATSM

INTERVENTIONS:
Drug: Cu(II)ATSM — copper-containing synthetic small molecule
  Other Names: diacetylbis(N(4)-methylthiosemicarbazonato) copper(II)

SUMMARY:
Multicenter, open-label dose-escalation study

DETAILED DESCRIPTION:
Multicenter, open-label, phase 1 study of Cu(II)ATSM administered orally to patients with early idiopathic Parkinson's disease. The study will be conducted in two phases. In the first phase, dose cohorts of six patients each will receive escalating daily doses of Cu(II)ATSM to establish the recommended phase 2 dose (RP2D). The starting dose will be 12 mg/day, which has been shown to be well tolerated in an ongoing phase 1 pharmacokinetic and dose-finding study of Cu(II)ATSM in patients with ALS (ClinicalTrials.gov identifier NCT02870634). In the second phase of the study, an expansion cohort of 20 patients will be treated at the RP2D to confirm tolerability and assess preliminary evidence of efficacy.

In both the dose escalation and expansion cohorts, once the first 28 days of treatment are completed, at the discretion of the investigator a patient may continue to receive Cu(II)ATSM treatment for a maximum of six 28-day treatment cycles.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent prior to initiation of any study-specific procedures
* Early idiopathic Parkinson's disease (PD) with at least two of the cardinal signs of PD (resting tremor, bradykinesia, rigidity, postural instability). If tremor is not present, must have unilateral onset and persistent asymmetry of symptoms.
* Hoehn & Yahr stage ≤ 2
* First PD motor symptoms occurred ≤ 5 years prior to screening visit
* Use of dopaminergic therapy allowed provided dose is stable for at least 8 weeks prior to screening visit
* Use of amantadine and/or anticholinergics allowed provided dose is stable for at least 8 weeks prior to screening visit
* Use of CNS-acting medications allowed provided dose is stable for at least 4 weeks prior to screening visit
* Age ≥ 30 years at time of PD diagnosis
* Adequate bone marrow reserve, liver and renal function:

Absolute neutrophil count ≥ 1500/µL; Platelet count ≥ 150,000/µL; Hemoglobin ≥ 11 g/dL; Creatinine clearance ≥ 6- mL/min (Cockroft & Gault formula); ALT and/or AST ≤ 2 x ULN; total bilirubin ≤ 1.5 x ULN; albumin ≥ 2.8 g/dL

* Women and men with partners of childbearing potential must take effective contraception while on study and women of childbearing potential must have a negative pregnancy test and be non-lactating at screening

Exclusion Criteria:

* Atypical Parkinsonism
* Taking ≥ 3 dopaminergic medications
* Exposure to typical or atypical antipsychotics or other dopamine blocking agents within 6 months prior to screening visit
* Exposure to any other investigational agent within 6 months or 2 investigational agents within 12 months prior to screening visit
* Known immune compromising illness or treatment
* History of brain surgery for PD, including deep brain stimulation and stem cell transplants
* History of cognitive or neuropsychiatric conditions
* Inability to swallow oral medications or presence of a GI disorder (eg, malabsorption) deemed to jeopardize intestinal absorption of study drug
* Active GI disease (excluding GERD) within 30 days prior to screening visit
* Presence of any of the following clinical conditions:

any significant non-PD CNS disorder; drug abuse or alcoholism; unstable cardiac, pulmonary, renal, hepatic, endocrine or hematologic disease; active infectious disease; AIDS or AIDS-related complex; malignancy within 3 years of screening (other than fully excised non-melanoma skin cancer, cured in situ cervical carcinoma, early stage bladder cancer, or DCIS of breast); psychosis or untreated major depression within 30 days of screening; dementia

* Current use of strong inducers or inhibitors of CYPs 2C19 and 2D6

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2017-08-14 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2020-02-29 (Actual)

PRIMARY OUTCOMES:
Recommended phase 2 dose | 6 months
  Recommended phase 2 dose as determined by the number of patients in each dose cohort with intolerance over up to six months treatment

SECONDARY OUTCOMES:
Treatment-related changes in disease severity | 6 months
  Treatment-related changes in disease severity assessed by the Unified Parkinson Disease Rating Scale (UPDRS)
Treatment-related changes in motor function | 6 months
  Treatment related changes in motor function assessed by the UPDRS Part III score and UPDRS ambulatory capacity subscore
Treatment-related changes in cognitive function | 6 months
  Treatment related changes in cognitive function assessed by the Montreal Cognitive Assessments (MoCA)
Treatment-related changes in quality of life | 6 months
  Treatment related changes in quality of life assessed by the 39-item Parkinson Disease Questionnaire (PDQ-39)
Treatment-related changes in constipation | 6 months
  Treatment related changes in constipation assessed by the Wexler Constipation Score

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Evans, MD, Principal Investigator — Melbourne Health
Locations (2):
- Australia (2):
  - Macquarie University, Macquarie Park, New South Wales
  - The Royal Melbourne Hospital, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: Yes
Plan to publish trial results and post results on www.ClinicalTrials.gov